CLINICAL TRIAL: NCT02926989
Title: Fluid Therapy in Acutely Ill Children - a Randomized Controlled Trial
Brief Title: Intravenous Fluids in Hospitalised Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: Oulu University Hospital (Other)
Responsible Party: Principal Investigator, Terhi Tapiainen, Adjunct professor, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EETTMK 48/2016
Record Dates: First submitted 2016-10-04; First posted 2016-10-06 (Estimated); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Hypokalemia; Hyponatremia; Hypernatremia; Dehydration
Keywords: Isotonic; Hypotonic; Intravenous fluids
MeSH Terms: conditions — Hypokalemia; Hyponatremia; Hypernatremia; Dehydration | interventions — Sodium Chloride; Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Isotonic solution (Experimental): Plasmalyte Glucos 50 mg/mL; total daily fluid requirements are estimated using the Holiday-Segar method plus possible dehydration (according to child's weight loss during acute illness); intravenous fluids are administered using delivery pumps programmed for an hourly infusion rate (mL/hour); intravenous fluids are administered as long as needed during hospitalization, but no longer than seven days after admission.
  Interventions: Drug: Plasmalyte Glucos 50 mg/mL
- Hypotonic solution (Active Comparator): 0.45% saline in 5% dextrose; total daily fluid requirements are estimated using the Holiday-Segar method plus possible dehydration (according to child's weight loss during acute illness); intravenous fluids are administered using delivery pumps programmed for an hourly infusion rate (mL/hour); intravenous fluids are administered as long as needed during hospitalization, but no longer than seven days after admission.
  Interventions: Drug: 0.45% saline in 5% dextrose

INTERVENTIONS:
Drug: Plasmalyte Glucos 50 mg/mL — Solution contains potassium chloride 5 mmol/L and sodium chloride 140 mmol/L.
  Other Names: ATC-code: B05BB02
  Arms: Isotonic solution
Drug: 0.45% saline in 5% dextrose — Solution contains potassium chloride 20 mmol/L and sodium chloride 80 mmol/L.
  Other Names: 0.45% NaCl in 5% dextrose.
  Arms: Hypotonic solution

SUMMARY:
The main objective of the trial is to evaluate the risk of hypokalemia following administration of a isotonic solution compared to a hypotonic solution in acutely ill hospitalised children, who need intravenous fluid therapy.

DETAILED DESCRIPTION:
The main objective of the trial is to evaluate the risk of hypokalemia (low plasma potassium concentration) following administration of a Plasmalyte Glucos 50 mg/mL solution compared to a 0.45% saline in 5% dextrose solution in acutely ill hospitalised children, who need intravenous fluid therapy. The secondary objective of the trial is to evaluate the risk of hyponatremia (low plasma sodium concentration) and the risk of hypernatremia (high plasma sodium concentration) following administration of isotonic solution compared to hypotonic solution.

ELIGIBILITY:
Inclusion Criteria:

* Acutely ill hospitalised children
* Need for intravenous fluid therapy

Exclusion Criteria:

* An initial plasma sodium concentration of lower than 130 mmol/L
* An initial plasma sodium concentration of higher than 150 mmol/L
* An initial plasma potassium concentration of lower than 3.0 mmol/L
* Need for 10% glucose solution
* Diabetes
* Diabetes insipidus
* Diabetic ketoacidosis
* Renal disease that needs dialysis
* Protocol-determined chemotherapy hydration
* Severe liver disease
* Inborn errors of metabolism that need protocol-determined fluid therapy

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 660 (Actual)
Dates: Start 2016-10-03 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Proportion of children with a clinically significant electrolyte disorder | Plasma sodium and potassium concentrations are assessed daily (at 7 am) during the intravenous fluid therapy from randomization up to seven days.
  Plasma potassium concentration<3.5 mmol/L, or hypernatremia >148 mmol/L, or hyponatremia <132 mmol/L

SECONDARY OUTCOMES:
Proportion of children with hyponatremia | Plasma sodium and potassium concentrations are assessed daily (at 7 am) during the intravenous fluid therapy from randomization up to seven days.
  Plasma sodium concentration of lower than 132 mmol/L.
Proportion of children with hypernatremia | Plasma sodium and potassium concentrations are assessed daily (at 7 am) during the intravenous fluid therapy from randomization up to seven days.
  Plasma sodium concentration of higher than 148 mmol/L.
Proportion of children with hypokalemia | 0-7 days from study entry
  Potassium < 3.5 mmol/L
Proportion of children with severe hypokalemia | 0-7 days from study entry
  Hypokalemia defined as concentration of potassium <3.0 mmol/L
Fluid retention (g) measured by the weight change | 0-7 days: Body weight is measured daily (at 7 am) during the intravenous fluid therapy from randomization up to seven days.
  Weight (g) at discharge - weight (g) at admission
Concentration of copeptin in plasma samples | 6-24 hours after study entry
  Copeptin plasma concentration
Concentration of bicarbonate (HCO3) in plasma samples | 1-3 days after study entry
  Plasma concentration of bicarbonate HCO3
Acidosis measured by pH in blood gas analysis | 1-3 days after study entry
  pH in the blood gas analysis
Alkalosis measured by base excess (BE) in blood gas analysis | 1-3 days after study entry
  Base excess in the blood gas analysis
Duration of intravenous fluid therapy | From randomization up to seven days.
  Hours from study entry to the stop of fluid therapy
Proportion of children who needed change of the study fluid treatment | From randomization up to seven days.
  Any change of the fluid used in the treatment
Proportion of children admitted to ICU | From randomization up to seven days.
  Admission to ICU for any reason
Time to discharge from hospital in hours | From randomization up to seven days.
  Time from study entry to discharge in hours
Number of deaths | 0-30 days from study entry
  Any death during the study

CONTACTS AND LOCATIONS:
Overall Officials: Terhi Tapiainen, MD, Principal Investigator — Oulu University Hospital
Locations (1):
- Oulu University Hospital, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lehtiranta S, Honkila M, Kallio M, Paalanne N, Peltoniemi O, Pokka T, Renko M, Tapiainen T. Risk of Electrolyte Disorders in Acutely Ill Children Receiving Commercially Available Plasmalike Isotonic Fluids: A Randomized Clinical Trial. JAMA Pediatr. 2021 Jan 1;175(1):28-35. doi: 10.1001/jamapediatrics.2020.3383. PMID 33104176